CLINICAL TRIAL: NCT07105124
Title: A Randomized, Open-label, Phase 1 Trial to Assess the Pharmacokinetics, Safety and Tolerability, and Pharmacodynamics of Sibeprenlimab Solution Administered Subcutaneously in Chinese Healthy Subjects
Brief Title: Safety and Tolerability, and PK of Sibeprenlimab in Chinese Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 417-201-00005
Record Dates: First submitted 2025-04-24; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects (HS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 200mg Sibeprenlimab (Experimental): 200 mg Sibeprenlimab (1 × 1 mL injection)
  Interventions: Drug: Sibeprenlimab
- 400mg Sibeprenlimab (Experimental): 400 mg Sibeprenlimab (1 × 2 mL injection)
  Interventions: Drug: Sibeprenlimab
- 600 mg Sibenlimab (Experimental): 600 mg Sibenlimab (1 × 1 mL injection and 1 × 2 mL injection)
  Interventions: Drug: Sibeprenlimab

INTERVENTIONS:
Drug: Sibeprenlimab — Sibeprenlimab is being developed for the treatment of immunoglobulin A nephropathy (IgAN), an autoimmune glomerulonephritis characterized by the deposition of immunoglobulin (Ig) A-containing immune complexes in the kidney.

SUMMARY:
A Trial to Assess the Pharmacokinetics, Safety and Tolerability, and Pharmacodynamics, of Sibeprenlimab Solution Administered Subcutaneously in Chinese Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Chinese subject between 18 and 55 years of age, inclusive, at the screening visit.
* Healthy, as determined by pretrial medical evaluation (medical history, physical examination, vital signs, 12-lead electrocardiogram [ECG], and clinical aboratory evaluations), as judged by the investigator.
* Body mass index between 19 and 32 kg/m2, inclusive, and body weight not less than 50 kg at the screening visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Screening clinical laboratory test values for IgA, IgG, and IgM must meet the following criteria (the clinical laboratory tests may be repeated once per the discretion of the investigator):

  * Serum IgA: ≥ 0.8 g/L
  * Serum IgG: ≥ 7.0 g/L
  * Serum IgM: ≥ 0.4 g/L

Exclusion Criteria:

* Subjects with potential to contribute to pregnancy who do not agree to practice 2 different approved methods of birth control or remain fully abstinent (periodic abstinence [eg, calendar, ovulation, symptothermal, post ovulation methods] or withdrawal are not acceptable methods of contraception) from the time of consent through the end of the subject's participation in the trial and an additional 90 days (biological male subjects) or 30 days (biological female subjects) thereafter. If employing birth control, 2 of the following methods must be used: vasectomy, tubal ligation, intrauterine device, birth control pill, birth control implant, birth control depot injection, birth control patch, condom with spermicide, sponge with spermicide, or occlusive cap (vaginal diaphragm or cervical/vault cap) with spermicide.
* Subjects must also agree not to donate sperm from the time of consent through the end of the subject's participation in the trial and an additional 90 days thereafter.
* Subject has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, blood dyscrasias or other medical disorder, including psychiatric disorders, cirrhosis, or malignancy. History of minor skin cancers (not including melanoma) or surgically treated, limited cervical carcinomas (ie, carcinoma in situ) are not exclusionary.
* History of a previous severe allergic reaction with generalized urticaria; angioedema or anaphylaxis.
* Known hypoglobulinemia disorder (ie, common variable immunodeficiency), X-linked agammaglobulinemia, selective IgA deficiency, selective IgM deficiency).
* History of chronic infection (eg, tuberculosis, osteomyelitis, etc) or any infection requiring hospitalization or treatment with antivirals, antibiotics, or antifungal therapy within 30 days prior to administration of IMP.
* Received vaccination during the 30 days prior to administration of IMP.
* Known hepatic (ie, prior or chronic hepatitis C or hepatitis B infection, nonalcoholic steatohepatitis, or cirrhosis) or biliary abnormalities (Gilberts syndrome or asymptomatic gallstones are permitted exceptions).
* A QT interval corrected for heart rate using Fridericia's correction (QTcF) > 450 msec for biological male subjects or > 470 msec for biological female subjects (may be repeated once).
* Previous receipt of antibody or biologic therapy whether licensed or investigational (Ig products, monoclonal antibodies, or antibody fragments) within 30 days prior to dosing or 5 half-lives within the dose of IMP, whichever is longer.
* Concomitant use of marketed or investigational system is immunosuppressive or immunomodulatory medications (eg, corticosteroids, methotrexate, azathioprine, etc. and/or biologics) is prohibited and require a washout period prior to screening (30 days or 5 half-lives, whichever is longer).
* Has received any prescription or nonprescription (over-the-counter [OTC]) medication during the last 30 days or 5 half-lives (of the drug in question), whichever is longer, preceding baseline (Day -1), with the exception of acetaminophen, ibuprofen (or an equivalent nonsteroidal anti-inflammatory drug), hormonal contraceptives, topical medications, vitamins, minerals, traditional Chinese medicines, and dietary or herbal remedies.
* Is participating in another clinical trial of any investigational drug, device, or intervention or has received any investigational medication during the last 3 months or 5 half-lives, whichever is longer, prior to the start of screening.
* History of or current hepatitis or acquired immunodeficiency syndrome or carriers of hepatitis B surface antigen, hepatitis C antibodies, and/or human immunodeficiency virus (HIV) antibodies.
* Subject with a positive drug or alcohol screen test result at screening or Day -1. The drug screen may be repeated once per the discretion of the investigator. The drug screen also screens for cannabinoids, methylenedioxymethamphetamine, and propoxyphene. If a subject tests positive on these tests, inclusion of that subject into the trial will be based on the investigator's judgment with consultation, as needed, with the medical monitor and the sponsor.
* Subject who has a history of alcohol or drug/chemical abuse.
* Subject who has donated > 500 mL or blood within 3 months prior to the start of screening.
* Subject who has donated any plasma within 7 days prior to baseline (Day -1).
* Is an employee of the clinical research team (any sponsor or trial site employee), or has a family member who is an employee of these organizations.
* Subject is judged by the investigator or the medical monitor to be inappropriate for the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Sibeprenlimab serum concentrations | Day 1 (predose, 4 hours postdose, and 8 hours postdose) and on Day 2 (24 hours postdose). All subjects will also have blood samples collected for PK analysis on Days 3, 5, 7, 9, 14 (Week 2), 28 (Week 4), 42 (Week 6), 56 (Week 8), 70 (Week 10), and 84
  Sibeprenlimab serum concentrations will be listed for each subject. Summary statistics of sibeprenlimab serum concentrations will be presented by dose level. Individual and mean sibeprenlimab concentration-time profiles will be plotted for each dose level in both linear and logarithmic scales.
  The following PK parameters for sibeprenlimab will be determined, as appropriate:
  Cmax AUC0-t AUC0-inf tmax t1/2,z CL/F

SECONDARY OUTCOMES:
total serum IgA | from 1st dose to day 84
  To characterize the effect of sibeprenlimab on total IgA

OTHER OUTCOMES:
IgG | Day 1 to Day 84
  Change from baseline in total serum IgG and IgM concerntrations and time to recovery
IgM | Day 1 to Day 84
  Change from baseline in total serum IgG and IgM concerntrations and time to recovery
APRIL | Day 1 to Day 84
  Changes in serum APRIL levels
ADA | Day 1 to Day 84
  Assess ADA status impact on sibeprenlimab PK parameters. Characterization of ADA levels Assess ADA status impact on sibeprenlimab PK parameters

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No